CLINICAL TRIAL: NCT05043701
Title: Individualized Systems Medicine Strategy for Targeting Cancer Stem Cells in Patients With Recurrent Glioblastoma (ISM-GBM)
Brief Title: Individualized Systems Medicine Functional Profiling for Recurrent Glioblastoma
Acronym: ISM-GBM
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Institute for Molecular Medicine (Other)
Responsible Party: Principal Investigator, Einar Vik-Mo, Head of Surgical Neuro-Oncology, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISM-GBM
Record Dates: First submitted 2021-06-07; First posted 2021-09-14 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Recurrent Glioblastoma
Keywords: functional screening; personalized treatment
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Intervention Model Description: Open labelled intervention study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Patients will be treated with drugs based on functional profiling of autologous tumor cells in vitro
  Interventions: Drug: Personalized drug combination

INTERVENTIONS:
Drug: Personalized drug combination — A personalized drug combination will be prescribed to each patient based on the functional drug screen

SUMMARY:
A study to determine the feasibility and safety of individualized cancer stem cell targeted therapy based on high-throughput functional profiling of FDA/EMA-approved drugs in patients with GBM that has recurred or progressed following standards-of-care (RT, TMZ).

DETAILED DESCRIPTION:
This protocol describes a prospective single-center phase 1 study to evaluate the feasibility and safety of a high-throughput drug sensitivity and resistance testing (HTS) platform of individualized cancer stem cells (CSC) to predict targeted therapies in patients with recurrence of GBM after standards-of-care. Secondary outcome include efficacy of drug treatment. The underlying hypotheses is that treatment of patients based on functional profiling og autologous CSCs using HTS a) is feasible within an acceptable time window for clinical translation, b) safely delay disease progression and c) increase survival. There are increasingly published literature that strongly support the importance of a targeting CSC to improve therapy and prevent tumor recurrence in GBM, as an additional strategy to improve the overall prognosis of patients.

ELIGIBILITY:
Inclusion Criteria:

* Recurrence of histologically verified glioblastoma
* Adequate biopsy to generate enough live cells to allow functional screening
* Must be ambulatory with an Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Must be 18 to 70 years of age
* Adequate bone marrow, liver and heart function
* Must be competent to give consent
* Signed informed consent and expected cooperation of the patients for the treatment and follow up must be obtained and documented according to International Conference on Harmonization Good Clinical Practice guidelines (ICH GCP), and national/local regulations.

Exclusion Criteria:

* Patients taking part in other clinical trials which could make inclusion or follow-up difficult
* Any reason why, in the opinion of the investigator, the patient should not participate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Drug screen completion and treatment initiation | 8 weeks after surgery
  The fraction of patient that can receive an individualized treatment based on drug screening. These drugs must be available for treatment and with a combined acceptable toxicity.

SECONDARY OUTCOMES:
Tumor response | 15 months from inclusion
  Tumor response by the chosen drug combination evaluated according to the updated response assessment in neuro-oncology (RANO) criteria.
Number of grade 3-5 adverse events | 15 months from inclusion
  Adverse events induced by selected treatments according to NCI Common Terminology Criteria for Adverse Events.
Overall survival | 15 months from inclusion
  Overall survival in treated patients from time of second surgery to all-cause mortality.
Patient reported quality of life, overall (QLQ-C30) | 15 months from inclusion
  Evaluated by Eastern Cooperative Oncology Group Quality of Life Questionaire (QLQ-C30), a questionnaire developed to assess the quality of life of cancer patients. Scale 30 to 120 points, where higher is worse.
Patient reported quality of life, brain specific(QLQ-BN20) | 15 months from inclusion
  Evaluated by Eastern Cooperative Oncology Group Quality of Life Questionaire, Brain module (QLQ-BN20). The brain cancer module is meant for use among brain cancer patients varying in disease stage and treatment modality. Scale 20 to 80 points, where higher is worse.

CONTACTS AND LOCATIONS:
Overall Officials: Einar O. Vik-Mo, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
Anonymized data will regarding tumor characteristics and results of functional profiling will be made available after publishing.

REFERENCES:
- [Background] Skaga E, Kulesskiy E, Brynjulvsen M, Sandberg CJ, Potdar S, Langmoen IA, Laakso A, Gaal-Paavola E, Perola M, Wennerberg K, Vik-Mo EO. Feasibility study of using high-throughput drug sensitivity testing to target recurrent glioblastoma stem cells for individualized treatment. Clin Transl Med. 2019 Dec 30;8(1):33. doi: 10.1186/s40169-019-0253-6. PMID 31889236
- [Background] Skaga E, Kulesskiy E, Fayzullin A, Sandberg CJ, Potdar S, Kyttala A, Langmoen IA, Laakso A, Gaal-Paavola E, Perola M, Wennerberg K, Vik-Mo EO. Intertumoral heterogeneity in patient-specific drug sensitivities in treatment-naive glioblastoma. BMC Cancer. 2019 Jun 25;19(1):628. doi: 10.1186/s12885-019-5861-4. PMID 31238897